CLINICAL TRIAL: NCT01331174
Title: Pulsed Short Wave in Females With Knee Osteoarthritis: A Multicenter, Randomized, Placebo-controlled Clinical Trial
Brief Title: Pulsed Short Wave in Females With Knee Osteoarthritis
Acronym: PSW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Irmandade da Santa Casa de Misericordia de Sao Paulo (Other)
Responsible Party: Principal Investigator, Thiago Yukio Fukuda, PhD, Irmandade da Santa Casa de Misericordia de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 403/06
Record Dates: First submitted 2011-04-05; First posted 2011-04-07 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Chronic Diseases; Knee Osteoarthritis
Keywords: knee; osteoarthritis; physical therapy; pulsed short wave
MeSH Terms: conditions — Chronic Disease; Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High dose PSW groups (Experimental): The treatment was performed with 2 devices named Diatermed II (Carci, São Paulo, SP, Brazil), previously calibrated, carrying frequency of 27.12MHz, peak power of 250W, and pulse duration of 400µs. All these parameters are predetermined in the device according to the manufacturer. We used the maximum power provided by the machine in a pulsed form with a pulse frequency of 145Hz, resulting in a mean power of 14.5W. These settings were based on the fact that applications with mean power below 20W minimize the thermal effects
  Interventions: Device: Pulsed short wave
- Placebo (Placebo Comparator): A placebo group was also established, in which the PSW device was turned on but kept in stand-by mode during 19 minutes without any electrical current being applied in the patients
  Interventions: Device: Pulsed short wave
- Control (No Intervention): The control group was composed of patients that were not submitted to any form of treatment and all patients were instructed to maintain their daily activities

INTERVENTIONS:
Device: Pulsed short wave — The treatment was performed with 2 devices named Diatermed II (Carci, São Paulo, SP, Brazil), previously calibrated, carrying frequency of 27.12MHz, peak power of 250W, and pulse duration of 400µs. All these parameters are predetermined in the device according to the manufacturer. We used the maximum power provided by the machine in a pulsed form with a pulse frequency of 145Hz, resulting in a mean power of 14.5W.
  Arms: High dose PSW groups; Placebo

SUMMARY:
Study design: Randomized clinical trial. Objective: To evaluate the effect of PSW treatment in different doses and to compare to the control and placebo group.

Background: Several forms of conservative treatment have been the focus of many recent studies in knee osteoarthritis (OA). Among these techniques, the application of pulsed short wave has been widely used, but the optimal dose and application time still have not been well established.

DETAILED DESCRIPTION:
Methods: One hundred and twenty-one females (average ± sd age, 60 ± 9 years), with a diagnosis of knee OA were distributed randomly into 4 groups: 35 patients who did not receive any treatment (control), 23 patients in the placebo group, 32 patients in the low dose PSW group (14.5W, 19 minutes and 17KJ), and 31 patients in the high dose PSW group (14.5W, 38 minutes and 33KJ). An 11-point numerical pain rating scale (NPRS) and "Knee Osteoarthritis Outcome Score" (KOOS) were used to assess pain and function in 3 stages: initial evaluation (pre-treatment), immediately after post-treatment, and a 12-month follow up.

Results: The 4 groups were homogeneous prior to treatment with respect to demographics, pain, and functional scales data. We demonstrated the short-term effectiveness of the PSW at low or high doses in patients with knee OA. Both treatment groups showed significant improvement in pain and function when compared to the control and placebo groups (P<0.05). There were no differences between PSW doses, despite the fact that a low dose of PSW seems to be more effective in the long term.

Conclusion: The PSW is an effective method for pain relief, functionality, and quality of life improvement in females with knee osteoarthritis in the short-term. On the basis of our results, we recommend PSW application in the female population with knee OA. However, conclusions regarding the 12-month follow up should be analyzed carefully due to the high dropout rate.

ELIGIBILITY:
Inclusion Criteria:

* The female subjects were included if they were over 40 with knee primary grade II or III OA, based on Gupta et al radiographic criteria2, and joint or anterior knee pain for at least 3 months.

Exclusion Criteria:

* We excluded patients with a history of surgery or any invasive procedure of the affected knee, physical therapy for knee injuries or any medication that had changed in the last 3 months, other diseases changing function, and patients who presented any contraindication for PSW application, especially metallic implants, pacemakers, lack of sensitivity, or tumor.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2006-08; Primary Completion 2008-03 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Pain evaluation | 1 year follow up
  The patients were evaluated in 3 phases: initial evaluation (pre-treatment), immediately after post-treatment, and a 12-month follow up. An 11-point numerical pain rating scale (NPRS) was used to measure pain during the last 2 days, where 0 corresponded to "no pain" and 10 corresponded to "worst imaginable pain".

SECONDARY OUTCOMES:
Functional evaluation | 1 year follow up
  We applied a validated "Knee Osteoarthritis Outcome Score" (KOOS) as a functional evaluation.28,29 The KOOS is a specific questionnaire for patients with knee injuries and OA. It consists of 5 subscales: symptoms, daily activities, pain, recreational function, and quality of life. The answers are based on reports from the last week, where 0 corresponded to "functional impairment" with exacerbated symptoms and 100 corresponded to "normal function" without symptoms. Each subscale was normalized and analyzed individually

CONTACTS AND LOCATIONS:
Overall Officials: Thiago Y Fukuda, PhD, Principal Investigator — Irmandade da Santa Casa de Misericórdia de São Paulo

REFERENCES:
- [Result] Fukuda TY, Ovanessian V, Alves da Cunha R, Jacob Filho Z, Cazarini Jr C, Rienzo FA, Centini AA. Pulsed Short Wave Effect in Pain and Function in patients with Knee Osteoarthritis. JARCET. 2008; 8(3):189-98.
- [Derived] Fukuda TY, Alves da Cunha R, Fukuda VO, Rienzo FA, Cazarini C Jr, Carvalho Nde A, Centini AA. Pulsed shortwave treatment in women with knee osteoarthritis: a multicenter, randomized, placebo-controlled clinical trial. Phys Ther. 2011 Jul;91(7):1009-17. doi: 10.2522/ptj.20100306. Epub 2011 Jun 3. PMID 21642511